CLINICAL TRIAL: NCT02069522
Title: Healthy Term Infants Fed Milk-Based Formulas With A Supplemental Carotenoid
Brief Title: Healthy Term Infants Fed Milk-Based Formulas
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: interim analysis findings
Sponsor: Abbott Nutrition (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple
Other Study IDs: AL13
Record Dates: First submitted 2014-02-18; First posted 2014-02-24 (Estimated); Last update posted 2015-03-24 (Estimated); Status verified 2015-03

CONDITIONS: Infants

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard Milk-based Formula Containing Carotenoid (Active Comparator): milk-based ready to feed infant formula
  Interventions: Other: Standard Milk-based Formula Containing Carotenoid
- Investigational Milk-based Formula Containing Carotenoid (Experimental): investigational milk-based ready to feed infant formula
  Interventions: Other: Investigational Milk-based Formula Containing Carotenoid

INTERVENTIONS:
Other: Standard Milk-based Formula Containing Carotenoid — Fed ad libitum
  Arms: Standard Milk-based Formula Containing Carotenoid
Other: Investigational Milk-based Formula Containing Carotenoid — Fed ad libitum
  Arms: Investigational Milk-based Formula Containing Carotenoid

SUMMARY:
This is a prospective, double blind, crossover study in healthy infants randomized to one of two study formulas. The trial will consist of two 21 day study feeding periods separated by a study washout period.

ELIGIBILITY:
Inclusion Criteria:

* Infant is in good health
* Infant is a singleton from a full term birth with a gestational age of 37-42 weeks
* Infant's birth weight was > 2490 g (~5 lbs 8 oz)
* Infant is between 14 and 28 days of age
* Parent(s) confirm intention to feed their infant the study product(s) as the sole source of nutrition for the duration of the study
* Parent(s) confirm intention not to administer vitamin or mineral supplements, DHA and ARA supplements, solid foods/juices to their infant from enrollment through the duration of the study

Exclusion Criteria:

* An adverse maternal, fetal or infant medical history that has potential for effects on tolerance, growth, and/or development.
* Infants using medications (including OTC), home remedies, herbal preparations, probiotics or rehydration fluids that might affect gastrointestinal (GI) tolerance

Ages: 14 Days to 28 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 91 (Actual)
Dates: Start 2014-02; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Carotenoid Concentration | Change from Baseline to end of Study Period A (~21 Days)
  Plasma sample

SECONDARY OUTCOMES:
Carotenoid Concentration | Change from Baseline to end Study Periods A (~21 Days) and B (~21 Days)
  Plasma sample

CONTACTS AND LOCATIONS:
Overall Officials: John B Lasekan, PhD, CCRP, Study Chair — Abbott Nutrition
Locations (6):
- United States (6):
  - Tuscon Medical Center, Tuscon, Arizona
  - Northpoint Pediatrics, Indianapolis, Indiana
  - Midwest Children's Health Research Institute, Lincoln, Nebraska
  - MetroHealth Medical Center, Cleveland, Ohio
  - Dayton Clinical Research, Dayton, Ohio
  - Institute of Clinical Research, Mayfield Heights, Ohio